CLINICAL TRIAL: NCT04973007
Title: Evaluation of Liver MR With an Abbreviated Gadobenate Dimeglumine Hepatobiliary Phase Protocol in Comparison to Liver MR With Gadoxetate Disodium for the Detection of Hepatic Metastases
Brief Title: Comparison of Contrast Agents in Liver MR for the Detection of Hepatic Metastases
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bracco Diagnostics, Inc (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 19-1045.cc; P30CA046934 (NIH)
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Oligometastatic Disease; Liver Metastases; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — gadolinium ethoxybenzyl DTPA; gadobenic acid

STUDY DESIGN:
Intervention Model Description: This is a prospective study. The subjects will be randomized into two groups. Both groups will undergo two complete protocol liver MRs for known or suspected CRC metastasis, one exam with gadoxetate disodium and the other exam with gadobenate dimeglumine, within an interval of 3-10 days, but in opposite order, determined randomly. From the complete protocol liver MR with both contrast agents, an image set of abbreviated HBP protocol liver MR for each agent will be obtained (Fig.1).Two week-intervals will be placed between the evaluations of different image sets of a patient, and the images will be presented in a different random order to each evaluating radiologist. The schedule of random order of protocol liver MRs and presentation of images to radiologists will be determined by the project biostatistician.
Who Masked: Outcomes Assessor
Masking Description: We have attempted to mitigate any potential conflict of interest through randomization of the order of exams and blinding the image evaluators to contrast agents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gadoxetate disodium exam first (Active Comparator): The subjects will be randomized into two groups. Both groups will undergo two complete protocol liver MRs for known or suspected CRC metastasis, one exam with gadoxetate disodium and the other exam with gadobenate dimeglumine, within an interval of 3-10 days, but in opposite order, determined randomly.
  Interventions: Drug: Gadoxetate disodium; Drug: Gadobenate dimeglumine
- Gadobenate Dimeglumine exam first (Active Comparator): The subjects will be randomized into two groups. Both groups will undergo two complete protocol liver MRs for known or suspected CRC metastasis, one exam with gadoxetate disodium and the other exam with gadobenate dimeglumine, within an interval of 3-10 days, but in opposite order, determined randomly.
  Interventions: Drug: Gadoxetate disodium; Drug: Gadobenate dimeglumine

INTERVENTIONS:
Drug: Gadoxetate disodium — Gadoxetate disodium is now mainly used for the purpose of HBP liver MR imaging to save MR scanner time and total examination time.
  Other Names: Primovist; Eovist
Drug: Gadobenate dimeglumine — The most commonly used MR contrast agent in abdominal imaging is gadobenate dimeglumine, which has mainly the characteristics of an extracellular agent used for most indications of MR examinations.
  Other Names: MultiHance

SUMMARY:
If an abbreviated HBP protocol liver MR with gadobenate dimeglumine is shown clinically comparable to standard of care liver MR with gadoxetate disodium for detecting hepatic metastasis from colorectal cancer, its use will save time, cost, and patients' effort.

DETAILED DESCRIPTION:
The goal is to:

* Estimate and compare the diagnostic performance, including sensitivity, specificity, positive/negative predictive value, and area under the receiver operating characteristics (AUROC), of abbreviated protocol liver magnetic resonance (MR) with hepatobiliary phase (HBP) using gadobenate dimeglumine for detecting liver metastases, with 1) abbreviated protocol liver MR with HBP using gadoxetate disodium, 2) standard of care complete protocol liver MR using gadoxetate disodium, and 3) complete protocol liver MR using gadobenate dimeglumine.
* Estimate and compare quantitative measures of HBP images (liver enhancement ratio, lesion contrast to noise and signal to noise ratios [CNR and SNR]) for both gadobenate dimeglumine and gadoxetate disodium.
* Qualitatively assess the preference, or lack thereof, of radiologists regarding the images generated by abbreviated protocol liver MR with HBP using gadobenate dimeglumine versus abbreviated protocol liver MR with HBP using gadoxetate disodium.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients
* Age 18-80 years
* No prior treatment including surgery
* Prior imaging with suspected liver metastasis

Exclusion Criteria:

* Age < 18 years or > 80 years
* eGFR < 30 ml/min/1.73 m2
* Previous reaction to gadolinium contrast agents
* History of claustrophobia or movement disorders likely to impact image quality
* Non-MR safe implants or metallic foreign bodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic Performance of gadobenate dimeglumine | 1 month
  The primary performance diagnostic will be sensitivity, similar to the recently published retrospective study by Canellas et al. (2019). In addition to other diagnostic performance metrics of interest (e.g., specificity, AUROC), lesions will be analyzed descriptively in terms of number of metastases detected and lesion size.
Quantitative Measures of hepatobiliary phase images | 1 month
  Mixed effects regression models will again be used to compare the three outcomes between methods, accounting for correlated data. The specific link function of the regression models will depend on the distributional characteristics of each outcome (e.g., logit link for dichotomous outcomes; linear regression for continuously measured outcomes).
Preference of radiologists for the images generated by amHBP versus aeHBP | 1 month
  The quality of amHBP and aeHBP images will be assessed with ordinal response mixed effect models that include right/left image as a covariate. We will assess if there was any reader specific and/or general bias to prefer an image on the left or the right of a screen, regardless of the amHBP or aeHBP, and consider this when modeling the probability of preference of amHBP over aeHBP. We will estimate the relative probabilities of no-preference, amHBP preference, or aeHBP preference.

SECONDARY OUTCOMES:
Compare Sensitivity and Specificity, | 1 month
  The primary analysis will use pathology as the gold standard, if available, but will revert to long term imaging in the absence of pathology. To address the potential impact of this limitation, we will also conduct an exploratory analysis to compare the sensitivity and specificity of the imaging methods by each gold standard.
Test Validity of Imaging Methods | 1 month
  We will also conduct an exploratory analysis to test the validity of long term imaging as a gold standard against available pathology reports.
Compare Patient Time Associated with Imaging Method | 1 month
  In addition to analyses for the primary aims, additional analyses will be conducted to examine patient time associated with each imaging method; time metrics can be compared between imaging methods in absolute terms, but also proportionally to sensitivity.
Compare Cost Associated with Imaging Method | 1 month
  In addition to analyses for the primary aims, additional analyses will be conducted to examine cost associated with each imaging method; cost metrics can be compared between imaging methods in absolute terms, but also proportionally to sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Madhuripan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No